CLINICAL TRIAL: NCT06724939
Title: Clinical Evaluation of Self-Adhesive Bulk-Fil Hybrid Composite Restoration in Primary Molars
Brief Title: Clinical Evaluation of Self-Adhesive Bulk-Fil Hybrid Composite in Primary Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A06020822
Record Dates: First submitted 2024-11-29; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Occlual Caries; Proximal Caries
Keywords: Bulk-fill composite; self-adhesive bulk-fill composite; primary molars; restorative treatment; occlusal lesions; occluso-proximal lesions

STUDY DESIGN:
Intervention Model Description: The children will be randomly divided into 2 main groups according to the type of carious lesion:Group I occlusal lesions.Group II occluso-proximal lesions.
  Then the children will be randomly sub grouped according to the type of restorative materials that will be used:Group IA and group IIA with filtek 3M bulk-fill resin composite .Group IB and IIB with surefil one restorative materials
Who Masked: Outcomes Assessor
Masking Description: The operator was not blinded to the allocation of the material because of the distinct application approach for the restorative materials, which prohibited doing so. However, the participants(children) ,their caregivers, and the statistician were blinded to the restorative material used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 3M bulk-fill composite resin class I (Active Comparator): class I bulk-fill composite
  Interventions: Other: self-adhesive bulk-fill resin composite
- 3M bulk-fill compsite resin class II (Active Comparator): class I bulk-fill
  Interventions: Other: self-adhesive bulk-fill resin composite
- surefil one class I (Experimental): class I surefil one
  Interventions: Other: self-adhesive bulk-fill resin composite
- surefil one class II (Experimental): class II surefil one
  Interventions: Other: self-adhesive bulk-fill resin composite

INTERVENTIONS:
Other: self-adhesive bulk-fill resin composite — surefil one self-adhesive bulk-fill composite

SUMMARY:
This study will evaluate the clinical performance of self-adhesive bulk-fill composite resin in the restoration of occlusal and occluso-proximal lesions in primary molars with hypothesis that there is no difference in the clinical performance of self-adhesive bulk-fill composite and traditional bulk-fill composite with adhesive over one year observation period

DETAILED DESCRIPTION:
Protocol of clinical procedure:After psychological management and preparation of the child, local anesthesia was administered in order to prevent pain upon cavity preparation and maintain the child's cooperation. Involved teeth were isolated using a rubber dam (DuraDam, Klang, Selangor D.E.,Malaysia). All cavities were cleaned and prepared using a high speed carbide bur (#330, MANI Inc, Tokyo, Japan) under a constant copious water-cooling system using a high-speed contra-angled hand piece (Dentsply Sirona, York, PA, USA). All occlusal pits and fissures were included in the cavity design to standardize the preparations. A small sectional contoured metal matrix (TOR VM, Russia) was placed interproximally and fixed with a wedge.

At this point, the operator defined the restorative material to be used by opening the allocation envelope.The cavities were restored in each subgroup with restorative material according to the manufacture instructions as follow:

In subgroup IA and IIA(cotrol groups), a 37% phosphoric acid etchant (Scotchbond Universal Etchant, 3M, ESP) was applied for 15 seconds on the dentine and 30 seconds on the enamel ,followed by washing for 40 seconds with water and gently air dried. The adhesive system (Scotchbond Universal Adhesive, 3M, ESPE, St. Paul, MN, USA) was applied actively to the entire surface using a disposable bond brush, for 20 seconds. The adhesive was dispersed into a thin layer with a gentle stream of air for 5 seconds, followed by light curing for 10 seconds using an LED light-curing unit (BluePhase N, Ivoclar Vivadent AG) with an intensity of 1200 mW/cm². Cavities were filled with FiltekTM Bulk Fill (St. Paul, MN, USA), in one increment and light cured for 20 seconds on each surface of the tooth with the same curing unit.

In subgroup IB and IIB (study groups), The cavities were cleaned using an air-water spray, leaving a moist cavity surface. Surefil one activated capsules (Dentsply Sirona, Konstanz, Germany) were mixed for 10 seconds using a capsule mixer (4200-5000 rpm) following the manufacturer's instructions. The restorative material was promptly dispensed into the prepared cavity using a capsule extruder. The dispensing process began at the cavity's deepest area, with the tip kept close to the bottom. The tip was gradually withdrawn as the cavity was filled in bulk and contoured with a hand instrument.(Following this, the restoration was cured for 20 seconds on each surface of the tooth with the same curing unit.

After that ,the occlusion was checked using articulating paper (Bausch, Nashua, NH, USA). The restorations were finished using a yellow-coded finishing flame stone (MANI Inc., Tokyo, Japan).Final polishing was performed using polishing disks (Soflex, 3M ESPE, MN, USA) while keeping the restoration moist with water spray.

Clinical evaluation: The restorations were evaluated clinically and radiographically according to Modified United States Public Health Organization (USHPS) criteria measuring marginal adaption, surface roughness, anatomic form, postoperative sensitivity, recurrent caries, retention, color match and proximal contact. These items were ranked according to the scores: Alpha -ideal clinical situation; Bravo-clinically acceptable; Charlie-clinically unacceptable situation. The evaluation was done post restoration(baseline) and at follow-up periods of 3, 6, and 12 months

ELIGIBILITY:
Inclusion Criteria:

* • Children with bilateral simple occlusal or occluso-proximal caries in the lower second primary molars.

  * Generally healthy children with no systemic disease.
  * Cooperative children with a behavior rating of 3 or 4 according to the Frankl Behavior Rating Scale.

Exclusion Criteria:

* Pulp exposure or indication for endodontic treatment or extraction.
* Teeth with symptoms such as spontaneous pain, swelling, infection, fistulae, abscesses or tenderness on percussion.
* Parents who weren't available for periodic follow up.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-19 (Estimated)

PRIMARY OUTCOMES:
Modified United States Public Health Organization (USPHS) criteria for evaluation | one year follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Mahmoud Abd El-Razzak, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rathke A, Pfefferkorn F, McGuire MK, Heard RH, Seemann R. One-year clinical results of restorations using a novel self-adhesive resin-based bulk-fill restorative. Sci Rep. 2022 Mar 10;12(1):3934. doi: 10.1038/s41598-022-07965-z. PMID 35273277